CLINICAL TRIAL: NCT06239753
Title: The Effect of Dynamic Neuromuscular Stabilization Applied in the Second Trimester of Pregnancy on Pregnancy: A Randomized Controlled Study
Brief Title: The Impact of Dynamic Neuromuscular Stabilization on Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dondu Kurnaz (Other)
Responsible Party: Sponsor-Investigator, Dondu Kurnaz, Doctor Associate Professor, Lütfi Kırdar City Hospital
Organization: Lütfi Kırdar City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KLKŞH
Record Dates: First submitted 2023-12-21; First posted 2024-02-02 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Pregnant; Exercise
Keywords: Pregnancy; Stabilization; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The complete randomization technique will be used for participant allocation to groups. This will be conducted through the https://www.randomizer.org/ website. Three computer-generated randomization sequences will be applied on a one-to-one basis. It has been observed that some numbers are assigned to all three groups in this system. To manage this situation, for individuals matching the same number, the person corresponding to that number in the group where the number first appeared will be assigned, and the next person will be assigned to the next group with the first unassigned number.
  Opaque envelope method will be used for group allocation. The researcher conducting the intervention and collecting the data forms will not be blinded to the groups, but the researchers responsible for measuring pelvic floor muscles, conducting analyses, and writing the findings will be blinded to the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic Neuromuscular Stabilization Applied (Experimental): Intervention Group I will receive DNS (Dynamic Neuromuscular Stabilization) applications in the hospital, led by a physiotherapist, once a week for 10 weeks. During each session, participants will be instructed to perform the DNS exercises at home and take notes. They will receive reminders via short message service (SMS) to practice the exercises at home. The DNS application for pregnant women involves checking the breathing pattern before starting exercises in all sessions. Pregnant women will be instructed to breathe through the nose, and if they find it challenging to maintain nasal breathing, the Body Oxygen Level Test (BOLT) score will be measured. If the BOLT score is low, guidance will be provided on how to increase it by adjusting the breathing technique."
  Interventions: Behavioral: Dynamic Neuromuscular Stabilization
- Standard Prenatal Education Program Implementation (Experimental): The group will receive the standard prenatal education program, consisting of 5 sessions of general education and 2 sessions of standard pregnancy exercises and respiratory exercises, as part of the hospital's prenatal education program. The educational topics will include one-hour sessions on pregnancy and nutrition, postpartum care and family planning, baby care and infant massage, breastfeeding and lactation education, and first aid for infants, under the headings of childbirth and coping methods for labor pain
  Interventions: Behavioral: Standard Prenatal Education Program Implementation
- Control (No Intervention): The control group will consist of pregnant women attending routine examinations at the hospital's maternity clinic. As per hospital policy, routine breastfeeding education is provided after the 32nd week during regular prenatal check-ups at the hospital.

INTERVENTIONS:
Behavioral: Dynamic Neuromuscular Stabilization — Conducting routine pregnancy examinations. Measurement of pelvic floor muscle dimensions. Providing education through prenatal classes. Application of Dynamic Neuromuscular Stabilization (DNS).
  Arms: Dynamic Neuromuscular Stabilization Applied
Behavioral: Standard Prenatal Education Program Implementation — Conducting routine pregnancy examinations. Measurement of pelvic floor muscle dimensions. Providing education through prenatal classes.
  Arms: Standard Prenatal Education Program Implementation

SUMMARY:
The aim of this randomized controlled study is to determine the pregnancy and childbirth outcomes of using the DNS method to facilitate anatomical and physiological adaptations during pregnancy.

DETAILED DESCRIPTION:
During pregnancy, significant anatomical and physiological changes occur as the baby grows inside the uterus. As pregnancy progresses, body mass index increases, the uterus expands towards the abdominal cavity, and the woman's center of gravity shifts. This change in the center of gravity leads to a backward shift in the trunk, hyperextension of the knees, and the formation of lumbar lordosis, thoracic kyphosis, and pelvic curvature. The increased weight can cause pelvic floor collapse and weakness in pelvic floor muscles, leading to urinary incontinence, pelvic organ prolapse, fecal incontinence, sexual dysfunction, and pelvic pain.

Proper management of the body during this period can not only facilitate childbirth but also reduce potential problems that may arise during pregnancy. Exercises play a crucial role in managing the body correctly during pregnancy. Aerobic exercises, strength training, and specific Kegel exercises are commonly performed during pregnancy. However, despite the frequent occurrence of musculoskeletal and postural changes during pregnancy, it is observed that postural exercises to regulate these changes are not widely implemented. Studies have indicated that stabilization exercises are more effective than traditional strength exercises in reducing complaints during pregnancy.

There is a lack of sufficient research in the literature on core stabilization related to posture alignment during pregnancy. Core stabilization is defined as the ability to control the position and movement of the trunk on the pelvis to allow optimal force production, transfer, and movement of the extremities. It is essential to prevent excessive load on the pelvis, spine, and kinetic chain. When this system functions effectively, loads on the body are distributed evenly, reducing excess load on the joints of the kinetic chain. Core strength training primarily focuses on strengthening deep core muscles, especially the multifidus and transversus abdominis muscles, which may weaken during pregnancy. Current exercise programs for pregnant women include exercises targeting core muscles, such as Pilates, antigravity fitness, birth support belts, stability balls, and Dynamic Neuromuscular Stabilization (DNS). Although studies on the benefits of stabilization exercises during pregnancy are available in the literature, there is no specific research on the application of DNS during pregnancy.

DNS is a system that emphasizes coordination and strength, focusing on the overall harmony of the body and foundational stability. It is based on developmental kinesiology models. DNS encompasses motor patterns and programs that infants inherently possess, allowing them to develop ideal posture, functional joint centering, optimal respiration, and locomotor skills during ontogenesis. The main goal is to restore physiological movement patterns defined by developmental kinesiology DNS has been widely accepted in clinical practice as a method that provides balanced subcortical or reflexive core stabilization, coordinating diaphragm, transversus abdominis, internal oblique, multifidus, and pelvic floor coactivation with intra-abdominal pressure and coordinated activation of superficial abdominal muscles.

Understanding the physiological and anatomical adaptations during pregnancy is crucial for the pregnant woman to cope with the increased metabolic demands vital for the developing fetus and meet the requirements of childbirth. Recognizing pathological deviations in pregnant women and ensuring core stabilization using appropriate methods are essential to optimize outcomes for both the mother and the baby. In the context of critically ill pregnant women, the DNS method can be used effectively during pregnancy, taking into account that different modifications may be needed to optimize their treatment. Well-designed studies are needed to determine the effectiveness of the DNS method.

ELIGIBILITY:
Inclusion Criteria:

Primiparity

* Singleton Pregnancy
* Gestational Age Between 11-13 Weeks
* Age Between 20-35 Years
* Body Mass Index in the Range of 18-30
* Receiving Pregnancy Check-ups at the Hospital where the Research is Conducted

Exclusion Criteria:

* Presence of a heart condition affecting hemodynamics
* History of restrictive lung disease
* Multiple pregnancies
* Severe anemia
* Movement-restricting musculoskeletal system anomalies

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Measurements | Between the 11th and 36th weeks of pregnancy,
  Pelvic floor muscle measurements will be assessed by a specialist in obstetrics and gynecology using transperineal ultrasonography. The Voluson 730 Pro ultrasound device will be used for assessment. A standard bladder filling protocol will be implemented before measurements. For this, women will be instructed to drink 600-750 ml of water one hour before the evaluation and refrain from emptying their bladders until the end of the test. Women will be positioned on their backs with knees flexed at 60°, and a pillow will be placed under their head. The ultrasound transducer will be placed suprapubically in the caudo-posterior direction to visualize the posterior inferior aspect of the bladder in the transverse plane during the first rest period. A first marker will be placed at the base of the bladder during this resting period. Women will be asked to contract their pelvic floor muscles during the assessment. The ultrasound image will be frozen during this contraction, and a second marker
The Pittsburgh Sleep Quality Index | Between the 11th and 36th weeks of pregnancy,
  Assessing sleep quality over the past month, the PSQI consists of a total of 24 questions. The total score ranges from 0 to 21. A total score higher than 5 indicates poor sleep quality. The scale will be applied twice, for the first and last application.
State-Trait Anxiety Inventory | Between the 11th and 36th weeks of pregnancy,
  Aims to measure individuals' levels of state and trait anxiety. The scale consists of two subscales, each comprising 20 items. An increase in scores from the scale indicates a higher level of anxiety. The scale will be applied twice, for the first and last application. The total score obtained from the scale varies between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety. The average score level determined in the applications varies between 36 and 41.
Oswestry Skalası | Between the 11th and 36th weeks of pregnancy,
  The questionnaire related to lower back pain consisting of a total of 10 questions, each with 6 options. The scale assigns a minimum score of 0 and a maximum score of 5 to each question. The overall possible score ranges from 0 to 50. An increase in the total score collected from the questionnaire indicates a worsening of the pain condition. The scale will be applied twice, for the first and last application.
Multidimensional Scale of Perceived Social Support | Between the 11th and 36th weeks of pregnancy,
  The questionnaire based on the subjective evaluation of social support received from family, friends, and significant others in individuals' social environments. The questionnaire examines three dimensions: family, friends, and significant others, totaling 48 questions with four questions evaluating each dimension. Each item in the scale is rated on a 7-point Likert scale ranging from strongly disagree to strongly agree. Scores obtained from the three separate dimensions are summed to calculate subscale scores, and the total scale score is obtained by summing the scores from all subscales. Higher scores from both the scale and its subscales indicate a higher perceived level of social support. The scale will be applied twice, for the first and last application. The score that can be obtained from the scale varies between 7 and 84.
The Fatigue Severity Scale | Between the 11th and 36th weeks of pregnancy,
  The Fatigue Severity Scale (FSS) was developed by Krupp et al. in 1989. The scale consists of a total of 9 items, and each item is rated on a scale of 1-7 (1=strongly disagree, 7=strongly agree). The total score is obtained by dividing the sum of scores by the number of scale items. The possible total score ranges from 9 to 63, and when divided by the number of items, the lowest possible score is 1, while the highest is 7. A higher score indicates an increased level of fatigue. The scale will be applied twice, for the first and last application.
Pregnancy Weight Gain | Between the 11th and 36th weeks of pregnancy,
  The weight of the pregnant woman will be measured at her first application and at her last application using the scale currently used for pregnant women.

SECONDARY OUTCOMES:
Blood pressure arterial (mmHg) | Between the 11th and 36th weeks of pregnancy,
  Blood pressure will be measured at the pregnant woman's first application and at her last application using the blood pressure monitor currently used for pregnant women.
pulse rate measurements | Between the 11th and 36th weeks of pregnancy,
  During the initial visit and the final visit, pulse rate measurements will be manually performed by the attending healthcare personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Ünlügedik Sayın, Dr., Principal Investigator — KLKŞH; Sunahan Koyuncu, Ftrp, Study Chair — KLKŞH; Döndü Kurnaz, Study Director — KLKŞH; Deniz Akyıldız, Study Chair — Sütçü İmam Unıversity
Locations (1):
- Lütfi Kırdar Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All researchers will only access data within the scope of their respective roles.